CLINICAL TRIAL: NCT04468022
Title: Toric Trifocal IOL Treatment With High Astigmatism and Hyperopia vs SMILE Enhancement After Trifocal IOL Treatment With High Astigmatism and Hyperopia
Brief Title: Toric Trifocal IOL Treatment With High Astigmatism and Hyperopia vs SMILE Enhancement After Trifocal IOL Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology, Eye Hospital Pristina Kosovo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EyeHospitalPristina
Record Dates: First submitted 2020-06-29; First posted 2020-07-13 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Astigmatism High Both; Pseudophakia; Hyperopia
Keywords: RELEX SMILE; Trifocal IOL; Toric Trifocal IOL
MeSH Terms: conditions — Pseudophakia; Hyperopia

STUDY DESIGN:
Intervention Model Description: Two groups divided in 40 eyes
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toric Trifocal IOL (Active Comparator): Twenty patients (20) underwent Toric Trifocal IOL surgery (first group)
  Interventions: Procedure: Toric Trifocal IOL
- Toric Trifocal IOL RELEX SMILE (Active Comparator): Twenty patients (20) underwent Toric Trifocal IOL and RELEX SMILE surgery (second group)
  Interventions: Procedure: Toric Trifocal IOL

INTERVENTIONS:
Procedure: Toric Trifocal IOL — Interventions are performed using a standard technique of sutureless phacoemulsification. In all cases, topical anesthesia was administered and pharmacologic mydriasis was induced using a combination of tropicamide and phenylephrine (10.0%). A mean clear corneal microincision of 2.2 mm was made with a knife according to position of the preop highest K value of the patient. A paracentesis was made 60 degree to 80 degree, clockwise from the main incision, and the anterior chamber was filled with an ophthalmic viscoelastic (OVD) after phacoemulsification/lensectomy and removal of clear lens. The IOL was subsequently implanted through the main incision using the BLUEMIXS 180 injector (Carl Zeiss meditec, Jena, Germany) for trifocal IOL , VISCOJECTTM BIO injector for toric trifocal IOL and then the OVD was removed. Postoperative pharmacologic treatment is performed with the combination of antibiotic and steroidal anti-inflammatory drops
  Other Names: Zeiss Meditec

SUMMARY:
The aim of this study is to assess visual and refractive outcomes after Toric Trifocal lens implantation and visual outcomes after laser vision correction (LVC) - ReLex Smile to correct residual refraction after 6 months of Toric Trifocal (IOL) implantation.

DETAILED DESCRIPTION:
The current state of the art for the correction of aphakia and presbyopia after lens extraction and refractive lensectomy is the implantation of multifocal intraocular lenses (IOL). In this study, the trifocal IOL types AT LISA TRI 839MP and AT LISA TRI TORIC 939MP (Carl Zeiss Meditec, Germany) were assessed.

In this prospective non-randomized study patients with spherical hypermetropia of >4 D in combination with high astigmatism of >3.0 D were treated. The first group of 40 eyes of 20 patients underwent refractive lensectomy, followed by implantation of the diffractive trifocal IOL type AT LISA TRI 839MP (Carl Zeiss Meditec, Jena, Germany) and 6 months later SMILE surgery. In 40 eyes of 20 patients in the second group IOL type AT LISA TRI TORIC 939MP were implanted. All patients were adequately consulted preoperatively about this type of IOLs and they were verbally consented. The study is adherent to the tenets of the Declaration of Helsinki. All patient are between 20- 45 years old.

The current study demonstrates that both the non-toric and toric versions of the trifocal IOL evaluated here provide excellent functional vision to patients, with good distance, intermediate and near uncorrected VA, a wide range of vision and good contrast sensitivity.

Before SMILE,Yag-Laser capsulotomy should be performed on all patients, regardless of posterior capsule ossification, in pseudophakic patients with residual refraction. When the Yag-Laser is applied after the Smile, there will be a diopter change.

Relex Smile surgery in pseudophakic patients with trifocal IOL was safe, effective, and predictable in a large cohort of patients. It is noteworthy that the decision for a treatment strategy (toric IOL or non-toric IOL with SMILE in s second step) should be made carefully, to select the appropriate method for the patient. During phaco surgey the positions of incisions should be determined according to the angle of the highest K value of the patient. For high astigmatic patients, toric trifocal IOL is highly effective.

ELIGIBILITY:
Inclusion Criteria:

1. High spherical hypermetropia
2. Astigmatismus >2 D or higher
3. Amblyopia
4. Strabismus (accomodative esotropia)

Exclusion Criteria:

1. Glaucoma
2. Retinal detachment
3. Corneal disease
4. Macular degeneration
5. Advanced Retinopathy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Measure of visual and refractive outcome after Toric Trifocal lens implantation | 6 months
  Complete ocular examination

SECONDARY OUTCOMES:
Measure of LVC using ReLex Smile to correct residual refraction after 6 months of Toric Trifocal IOL | 6 months
  Complete ocular examination

OTHER OUTCOMES:
UDVA, CDVA, CNVA, Goldmann applanation tonometry | 6 months
  Examinations used

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Semiz, Dr., Principal Investigator — Principal Doctor
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04468022/Prot_SAP_000.pdf